CLINICAL TRIAL: NCT00483288
Title: Wake Forest University Cervical Screening and Follow Up System for Hispanic Women - A Pilot Study
Brief Title: Written Educational Information and Phone Calls in Increasing Follow-Up Care in Hispanic Women With Abnormal Pap Smears
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Health Services Research
Other Study IDs: CCCWFU-30104B; CDR0000547179 (Registry Identifier: PDQ (Physician Data Query)); CCCWFU-BG04-578
Record Dates: First submitted 2007-06-06; First posted 2007-06-07 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2013-06

CONDITIONS: Cervical Cancer
Keywords: cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Early Intervention, Educational

INTERVENTIONS:
Other: educational intervention
Other: questionnaire administration
Other: study of socioeconomic and demographic variables
Other: survey administration

SUMMARY:
RATIONALE: Written educational materials and counseling by phone may help promote follow-up care in women with abnormal Pap smears.

PURPOSE: This clinical trial is studying how well written educational information and phone calls work in increasing follow-up care in Hispanic women with abnormal Pap smears.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the reasons for nonadherence to follow-up in Hispanic women with abnormal Pap smear findings.
* Assess the effect of written educational information and phone calls on follow-up rate in these patients.

OUTLINE: This is a pilot, cross-sectional, controlled, multicenter study. Patients are sequentially assigned to 1 of 3 intervention groups.

* Group 1 (control): Patients complete a standardized Spanish survey questionnaire, assessing their demographic information, knowledge, attitudes, behaviors, experiences with cervical screening, past medical history, and prior treatment, either in person (for those who kept their colposcopy appointment) or over the telephone (for those who did not keep their colposcopy appointment). Additional questions are added for patients who did not keep their colposcopy appointment to test for differences and to learn the reasons for not keeping their appointment.
* Group 2 (written educational information): Patients receive notification of their colposcopy appointment and an educational letter about Pap smears, cervical cancer risk, and the purpose and procedure of colposcopy. They complete the standardized Spanish survey questionnaire as in group 1.
* Group 3 (phone call): Patients receive notification of their colposcopy appointment and a personal telephone call educating them about Pap smears, cervical cancer risk, and the purpose and procedure of colposcopy. They complete the standardized Spanish survey questionnaire as in group 1.

All patients are asked to agree to submit residual Pap smear fluid to the Comprehensive Cancer Center of Wake Forest University tumor bank, and be included in a tracking system to insure future follow-up communications.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Abnormal Pap smear findings indicating the need for further treatment at the colposcopy clinic
* Scheduled for colposcopy at the Comprehensive Cancer Center of Wake Forest University
* No history of invasive cervical cancer

PATIENT CHARACTERISTICS:

* Must be of Hispanic background, including any of the following:

  * Hispanic
  * Latino
  * Chicano
  * Mexican American
  * Puerto Rican
  * Cuban American

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2005-05; Primary Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Reasons for nonadherence to follow-up
Effect of written educational information and phone calls on follow-up rate

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte E. Miller, MD, Study Chair — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States